CLINICAL TRIAL: NCT02285907
Title: The Effects of Consuming Beef vs. Soy-rich Lunch Meals, Matched for Macronutrient Content or Serving Size, on Markers of Appetite Control and Satiety
Brief Title: Protein Quality on Appetite Control, Reward-driven Eating, & Subsequent Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Heather Leidy, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: UMissouri
Record Dates: First submitted 2014-10-24; First posted 2014-11-07 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Appetite and General Nutritional Disorders
MeSH Terms: interventions — Nutrients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Macronutrient and Fiber Matched BEEF (Experimental): The participants will consume the macronutrient and fiber matched BEEF lunch on a single testing day. BEEF contained 33% protein, 43% CHO, and 24% fat; the BEEF meal contained 24 g of beef protein from 96% lean ground beef (Cargill, KS). Soy fiber (Nutritional Designs, NY) was added to the BEEF meal to match total final content between meals.The participants will consume the serving size matched BEEF lunch on a single testing day. BEEF contained 33% protein, 43% CHO, and 24% fat; the BEEF meal contained 24 g of beef protein from 96% lean ground beef patty (Cargill, KS).
  Interventions: Other: Macronutrient and Fiber Matched BEEF
- Macronutrient and Fiber Matched SOY (Experimental): The participants will consume the macronutrient and fiber matched SOY lunch on a single testing day. SOY contained 33% protein, 43% CHO, and 24% fat; the SOY meal contained 24 g of textured soy protein concentrate (Boca Foods, WI).
  Interventions: Other: Macronutrient and Fiber Matched SOY
- Serving Size Matched BEEF (Experimental): The participants will consume the serving size matched BEEF lunch on a single testing day. BEEF contained 33% protein, 43% CHO, and 24% fat; the BEEF meal contained 24 g of beef protein from 96% lean ground beef patty (Cargill, KS).
  Interventions: Other: Serving Size Matched BEEF
- Serving Size Matched SOY (Experimental): The participants will consume the serving size matched SOY lunch on a single testing day. SOY contained 24% protein, 49% CHO, and 24% fat; the SOY meal contained 14 g of textured soy protein concentrate (Boca Foods, WI).
  Interventions: Other: Serving Size Matched SOY

INTERVENTIONS:
Other: Macronutrient and Fiber Matched BEEF — The participants will consume the macronutrient and fiber matched BEEF lunch on a single testing day. BEEF contained 33% protein, 43% CHO, and 24% fat; the BEEF meal contained 24 g of beef protein from 96% lean ground beef (Cargill, KS). Soy fiber (Nutritional Designs, NY) was added to the BEEF meal to match total final content between meals.The participants will consume the serving size matched BEEF lunch on a single testing day. BEEF contained 33% protein, 43% CHO, and 24% fat; the BEEF meal contained 24 g of beef protein from 96% lean ground beef patty (Cargill, KS).
  Arms: Macronutrient and Fiber Matched BEEF
Other: Macronutrient and Fiber Matched SOY — The participants will consume the macronutrient and fiber matched SOY lunch on a single testing day. SOY contained 33% protein, 43% CHO, and 24% fat; the SOY meal contained 24 g of textured soy protein concentrate (Boca Foods, WI).
  Arms: Macronutrient and Fiber Matched SOY
Other: Serving Size Matched BEEF — The participants will consume the serving size matched BEEF lunch on a single testing day. BEEF contained 33% protein, 43% CHO, and 24% fat; the BEEF meal contained 24 g of beef protein from 96% lean ground beef patty (Cargill, KS).
  Arms: Serving Size Matched BEEF
Other: Serving Size Matched SOY — The participants will consume the serving size matched SOY lunch on a single testing day. SOY contained 24% protein, 49% CHO, and 24% fat; the SOY meal contained 14 g of textured soy protein concentrate (Boca Foods, WI).
  Arms: Serving Size Matched SOY

SUMMARY:
To determine whether the consumption of a beef-rich lunch improves appetite control, satiety, and energy intake regulation while reducing food reward and food cravings compared to the consumption of a soy-rich lunch when matched for macronutrients and fiber content or when match for serving size. The mechanisms of action surrounding the differential responses of beef versus soy proteins were also explored.

DETAILED DESCRIPTION:
A randomized, crossover design, acute study was completed in 21 healthy adults (age 23 ±1 y; BMI: 23.8 ± 0.6 kg/m2) to compare 400 kcal lunch meals varying in protein quality. Two separate comparisons were performed. The first comparison consisted of macronutrient and fiber-matched lunches which varied in protein quality: 24 g beef protein vs. 24 g soy protein. The second comparison matched serving size only: 1 serving of beef (24 g protein with 0 g fiber) vs. 1 serving of soy (14 g protein; 5 g fiber). For each treatment, the participants completed 2 testing days per lunch treatment. During the "Appetite Assessment Days," each participant reported to the lab to consume one of the lunch meals. Pre and 7-h post-lunch appetite and cravings questionnaires were completed throughout each testing day along with plasma, hormonal responses, and plasma amino acid concentrations through repeated blood sampling. Ad libitum dinner energy intake was also measured. During the "Reward Assessment Days," the participants reported to our facility to again consume one of the lunch meals. Pre and post-lunch neural responses to food stimuli, through functional magnetic resonance imaging (fMRI), occurred followed by ad libitum consumption of a lunch dessert.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-30 y
* Normal to Overweight (BMI: 18-29.9 kg/m2)
* No metabolic, psychological, or neurological diseases/conditions
* Not currently/previously on a weight loss or other special diet (in the past 6 months)
* Not a vegetarian
* Right-handed (necessary for the fMRI analyses)
* Not pregnant
* Meets the MU-Brain Imaging Center Screening Criteria
* Have not given blood (for the American Red Cross in the past 6 months)

Exclusion Criteria:

* Age >30 y and <18y
* Under Weight or Obese (BMI: <18 kg/m2 or >29.9 kg/m2)
* Clinically diagnosed with diabetes (Type I or Type II), having an eating disorder, or having any other metabolic, psychological, or neurological diseases/conditions that would influence the study outcomes.
* Currently/previously on a weight loss or other special diet (in the past 6 months)
* Left-handed
* Claustrophobic (≥ 2 past bouts of claustrophobia when exposure to small spaces)
* Do not meet the fMRI criteria established by the MU-BIC (regarding metal implants, etc.)
* Pregnant
* Does not meeting the MU-Brain Imaging Center screening criteria
* Have given blood (for the American Red Cross) in the past 6 months or plan to give blood in the following 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Douglas SM, Lasley TR, Leidy HJ. Consuming Beef vs. Soy Protein Has Little Effect on Appetite, Satiety, and Food Intake in Healthy Adults. J Nutr. 2015 May;145(5):1010-6. doi: 10.3945/jn.114.206987. Epub 2015 Mar 25. PMID 25809680

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Twenty-four participants signed the consent but two withdrew prior to beginning testing day procedures. One participant was withdrawn due to protocol violations prior to beginning the fourth treatment. All 21 remaining participants completed all interventions of a randomized cross-over study to compare 400-kcal lunch meals varying in protein quality but matched for either macronutrient or fiber content or serving size (Macronutrient and Fiber Matched BEEF, Macronutrient and Fiber Matched SOY, Serving Size Matched BEEF, and Serving Size Matched Soy). The participants completed 2 testing days per lunch treatment. On the first day, participants completed the 8 hour testing day with repeated blood sampling and appetite questionnaires. During the second testing day, pre- and post-lunch food cue-stimulated fMRI brain scans were completed. Within each treatment, the first and second testing days were separated by 2-7 days. However, there was 7-14 days in between each treatment.
Period: Overall Study
Arm/Group | All Study Participants
Started | 21
Began 1st Intervention | 21
Began 2nd Intervention | 21
Began 3rd Intervention | 21
Began 4th Intervention | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All 21 participants completed all interventions of a randomized cross-over study to compare 400-kcal lunch meals varying in protein quality but matched for either macronutrient or fiber content or serving size. In the macronutrient and fiber-matched comparisons, both lunch meals contained 24-g protein and 2-g fiber, differing only in the type of protein consumed (beef vs. soy). In the serving size-matched comparisons, the lunch meals contained 1 serving of beef (24-g protein/1-g fiber) or 1 serving of soy (14-g protein/5-g fiber). The participants completed 2 testing days per lunch treatment. On the first day, participants completed the 8 hour testing day with repeated blood sampling and appetite questionnaires. During the second testing day, pre- and post-lunch food cue-stimulated fMRI brain scans were completed. Within each treatment, the first and second testing days were separated by 2-7 days. However, there was 7-14 days in between each treatment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Eating Initiation
Description: Eating initiation will be measured as the time lapse between consuming the intervention and requesting dinner.
Time Frame: 1 Day
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Macronutrient and Fiber Matched Beef | Macronutrient and Fiber Matched Soy | Serving Size Matched Beef | Serving Size Matched Soy
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | 250 (15) | 270 (20) | 245 (25) | 250 (20)

2. Primary Outcome: Subsequent Food Intake
Description: Ad libitum dinner and snacks were provided. Energy content and macronutrient content of these eating occasions were assessed.
Time Frame: 1 Day
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | Macronutrient and Fiber Matched Beef | Macronutrient and Fiber Matched Soy | Serving Size Matched Beef | Serving Size Matched Soy
Number analyzed (Participants) | 20 | 20 | 20 | 20
kilocalories | 240 (74) | 970 (82) | 920 (75) | 900 (72)

3. Primary Outcome: Net Incremental Area Under the Curve (niAUC) of Perceived Hunger and Fullness
Description: Computerized questionnaires, assessing perceived sensations of hunger and fullness were completed throughout the testing days. The questions are worded as "how strong is your feeling of" with anchors of "not at all" to "extremely." Each reported score can be a minimum of 0 and a maximum of 100 mm. niAUC was calculated for by computing the summation of the average change from baseline score (units of mm) for each time point and the subsequent time point, multiplied by the difference in time (min) between the two measures. For reported feelings of hunger, a higher score can be interpreted as "feeling more hungry." For fullness, higher can be interpreted as "feeling more full." Questionnaires were asked at baseline and about every 30 minutes throughout the day for a total of 20 questionnaires.
Time Frame: - 15 min, +0 min,+30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min, +255 min, +270 min, +285 min, +300 min, +330 min, +360 min, +390 min, +420 min, +450 min, and +480 min
Measure: Mean (Standard Error); unit: mm*min
Arm/Group | Macronutrient and Fiber Matched Beef | Macronutrient and Fiber Matched Soy | Serving Size Matched Beef | Serving Size Matched Soy
Number analyzed (Participants) | 20 | 20 | 20 | 20
mm*min
  "How strong is your feeling of hunger?" | 45 (1000) | -2840 (1650) | -1360 (1410) | 745 (1480)
  "How strong is your feeling of being full?" | 2440 (1360) | 3320 (1600) | 2270 (1220) | 1910 (1560)

4. Primary Outcome: Net Incremental Area Under the Curve (niAUC) of Plasma Total Glucagon-like Peptide (GLP-1) and Total Peptide YY (PYY)
Description: The samples were collected in test tubes containing ethylenediaminetetraacetic acid. Protease inhibitors (pefabloc SC and dipeptidyl peptidase) were added to some of the tubes to reduce protein degradation. The plasma was separated and stored at -80°C. Plasma total glucagon-like peptide (GLP-1) and peptide YY (PYY) were measured for all time points using the Milliplex multi-analyte profiling magnetic bead-based multi-analyte, metabolic panel, 2-plex assay and Magpix Luminex technologies. niAUC was calculated throughout the testing period by computing the summation of the average change from baseline score (units of pg/ml) for each time point and the subsequent time point, multiplied by the difference in time (units of min) between the two time instances for a total of 20 blood samples.
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: (pg*min)/ml
Arm/Group | Macronutrient and Fiber Matched Beef | Macronutrient and Fiber Matched Soy | Serving Size Matched Beef | Serving Size Matched Soy
Number analyzed (Participants) | 20 | 20 | 20 | 20
(pg*min)/ml
  GLP-1 | 4100 (811) | 2790 (1450) | 2120 (916) | 4870 (1200)
  PYY | 1590 (944) | 1330 (1710) | 1980 (1720) | 1720 (6430)

5. Primary Outcome: Food Cue-stimulate fMRI Brain Scans
Description: Participants viewed 3 categories of pictures including food, nonfood (animals), and blurred baseline images. The pictures from each category were presented in blocks of images. Animal pictures were used to control for visual richness and general interest (i.e., appealing but not appetizing). To determine the effects of protein type on neural activity associated with food motivation, repeated measures ANOVAs were performed on the brain activation maps within the Brain Voyager software with use of stimulus [food (i.e., appetizing and appealing) vs. nonfood (i.e., animal, nonappetizing but appealing] and protein source (BEEF vs. SOY) comparisons within the macronutrient and fiber-matched condition and the serving size-matched conditions, separately. The mean percent signal change in the maximum voxel within each region that displayed significant activation after the BEEF and SOY meals was then determined. Talairach coordinates for each region are presented for each row as (x;y;z).
Time Frame: 3 hours
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Serving Size Matched Beef | Serving Size Matched Soy
Number analyzed (Participants) | 21 | 21
percent signal change
  Post-Pre lunch Anterior Cingluate (2;25;0) | -22 (6) | 7 (9)
  Post-Pre lunch Insula (-40;10;-8) | -30 (6) | -7 (10)

6. Secondary Outcome: Plasma Amino Acids
Description: Plasma amino acid concentrations were measured from the pre and hourly postprandial time points until dinner request following the Macronutrient and Fiber Matched BEEF meal and the Serving Size Matched Beef Meal. An average amino acid concentration was then determined from the change from baseline concentration for all available time points. Plasma amino acid analyses were performed through the University of Missouri-Columbia Agricultural Experiment Station Chemical Laboratories using cation-exchange chromatography (cIEC-HPLC) coupled with post-column ninhydrin derivatization and quantitation.
Time Frame: as for outcome 3
Population: Four participants were excluded because of insufficient time points.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Macronutrient and Fiber Matched Beef | Serving Size Matched Beef
Number analyzed (Participants) | 17 | 17
pg/ml
  Taurine | 0.24 (0.18) | -0.78 (0.25)
  Valine | 4.01 (1.09) | 0.03 (0.86)
  Methionine | 0.64 (0.22) | 0.04 (0.18)
  Isolecuine | 2.51 (0.60) | 1.04 (0.38)
  Leucine | 4.68 (1.06) | 1.61 (0.65)
  Tyrosine | 1.49 (0.57) | 0.12 (0.35)
  Phenylalanine | 0.40 (0.34) | -0.13 (0.33)
  Tryptophan | 4.78 (0.41) | 2.65 (0.51)
  Lysine | 5.02 (1.26) | 0.33 (1.07)
  Histidine | 1.41 (0.44) | -0.29 (0.33)
  Tryptophan/Large Neutral Amino Acids | 0.020 (0.004) | 0.019 (0.005)
  Total Amino Acids | 29.13 (10.90) | -6.35 (8.63)

ADVERSE EVENTS:
Time Frame: Adverse data was collected from when they began study procedures to when the completed all testing procedures (approximately 1 month). The length of the study (beginning with the first participant and ending with the last participant) spanned approximately 7 months.
Groups:
- Macronutrient and Fiber Matched BEEF; Macronutrient and Fiber Matched SOY: The participants will consume the macronutrient and fiber matched SOY lunch on a single testing day. SOY contained 33% protein, 43% CHO, and 24% fat; the SOY meal contained 24 g of textured soy protein concentrate (Boca Foods, WI).
Arm/Group | Macronutrient and Fiber Matched BEEF | Macronutrient and Fiber Matched SOY | Serving Size Matched BEEF | Serving Size Matched SOY
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No